CLINICAL TRIAL: NCT03450837
Title: Diminished Macrophage Cholesterol Efflux Mediated by HDL and Coronary Artery Disease in Young Male Anabolic Androgenic Steroid Users
Brief Title: Impaired HDL and Coronary Artery Disease in Anabolic Androgenic Steroid Users
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria Janieire de Nazaré Nunes Alves, PhD, University of Sao Paulo General Hospital
Other Study IDs: CAD-AnabolicAndrogenicSteroids
Record Dates: First submitted 2018-02-15; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; HDL; anabolic steroids
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anabolic androgenic steroids users: This group had been involved in strength training for at least 2 years, self-administering anabolic androgenic steroids in periodic cycles lasting from 8 to 12 weeks for at least 2 years with 2-4 cycles per year. All participants were on a cycle over the course of the study.
  Coronary Computed Tomography Angiography and Macrophage cholesterol efflux mediated by HDL
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography; Diagnostic Test: Macrophage cholesterol efflux mediated by HDL
- Anabolic androgenic steroids nonusers: This group had been involved in strength training for at least 2 years and they have never took anabolic androgenic steroids.
  Coronary Computed Tomography Angiography and Macrophage cholesterol efflux mediated by HDL
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography; Diagnostic Test: Macrophage cholesterol efflux mediated by HDL
- Sedentary control: This group were sedentary men without cardiovascular disease.
  Coronary Computed Tomography Angiography and Macrophage cholesterol efflux mediated by HDL
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography; Diagnostic Test: Macrophage cholesterol efflux mediated by HDL

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomography Angiography — To assess coronary artery plaque and calcification, all participants underwent coronary computed tomography angiography according to the guidelines of the Society of Cardiovascular Computed Tomography (SCCT). All CT scans were acquired in a 320-row detector scanner (AquillionOneTM - Toshiba Medical Systems Corporation, Otawara, Japan) with 0.5-mm thick slices. Acquisition protocol included coronary artery calcium scoring (CACS) and coronary CTA. CACS protocol utilized a 370-ms tube rotation, 120-kV tube voltage, 300-mA tube current, and 320x0.5-mm collimation with 3-mm slice thickness reconstructed images, one heart beat acquisition during diastole.
Diagnostic Test: Macrophage cholesterol efflux mediated by HDL — Macrophages were incubated with DMEM (Low Glucose, Gibco, Grand Island, New York, USA) containing 1 mg fatty acid free albumin (FAFA) (Sigma-Aldrich, Steinheim, Germany) plus 50 μg acetylated LDL/mL and 0.3 μCi 14C-cholesterol/mL (Amersham Biosciences, UK) for 48h. After washing with PBS/FAFA, cells were incubated in the presence or absence of HDL (50 µg/mL) for 8h. The amount of radioactivity present in the medium at the end of the HDL incubation period will indicate albumin-mediated cholesterol efflux with albumin alone and total efflux with albumin + HDL. Thus, specific HDL-mediated efflux will be calculated, subtracting the albumin-mediated efflux from total efflux

SUMMARY:
Anabolic androgenic steroids (AASs) have been associated with coronary artery disease (CAD). The illicit use of these substances also leads to a remarkable decrease in high-density lipoprotein (HDL) plasma concentration, which could be a key factor in the atherosclerotic process. The investigators tested the functionality of HDL by cholesterol efflux and antioxidant capacity and its association with CAD in young men.

DETAILED DESCRIPTION:
Twenty strength-trained AAS users (AASU) age 29±5 yr, 20 age-matched strength-trained AAS nonusers (AASNU), and 10 sedentary controls (SC) were enrolled.

HDL concentration and functionality by measuring the 14C-cholesterol efflux mediated by HDL and the ability of HDL in inhibiting LDL oxidation were evaluated.

Coronary artery was evaluated with coronary computed tomography angiography.

ELIGIBILITY:
Inclusion Criteria:

* Anabolic androgenic steroids users and Anabolic androgenic steroids nonusers groups had been involved in strength training for at least 2 years;
* Anabolic androgenic steroids users should be self-administering anabolic androgenic steroids in periodic cycles lasting from 8 to 12 weeks for at least 2 years with 2-4 cycles per year;
* All anabolic androgenic steroids users were on a cycle over the course of the study;
* Sedentary control group: sedentary men without cardiovascular disease.

Exclusion Criteria:

* Smoking;
* Alcohol consumption;
* Use of diuretics and/or antihypertensive medications;
* Liver and kidney disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anabolic androgenic steroids users and nonusers were recreational weightlifters or amateur bodybuilding athletes who were recruited from gymnasiums.
  Sedentary control group was recruited from community sample.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Concentration and the functionality of HDL | 1 day
  Blood sample was collected in the morning (between 8:00-10:00 a.m.) after 12 hours fasting and after 30 minutes of resting for HDL concentration assessment.
  Determination of 14C-cholesterol efflux mediated by HDL utilized macrophages cultured cells from mice was used to test the functionality of HDL.

SECONDARY OUTCOMES:
Prevalence of CAD in young men anabolic steroids users | 1 day
  Coronary computed tomography angiography was used to evaluate coronary artery plaque and calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Janieire NN Alves, MD, Principal Investigator — Heart Institute

IPD SHARING:
Plan to Share IPD: No